CLINICAL TRIAL: NCT02530346
Title: Is Colostomy Closure Without Mechanical Bowel Preparation Safe in Pediatric Patients? Randomized Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Emilio Fernandez Portilla, Pediatric Colorectal Surgery Attending, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIM-2015-087
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Colostomy; Surgical Anastomosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mechanical Bowel Preparation (Active Comparator): Patients will receive enteric polyethylene glycol at 100 ml/kg/dose during 4 hours, and up to 3 times, prior to surgery.
  Enemas with normal saline 20 ml/kg/do will be administered through the stomas 3 times a day
  Interventions: Drug: Mechanical Bowel Preparation
- No Mechanical Bowel Preparation (Experimental): Patients will not receive any preparation prior to surgery
  Interventions: Drug: No Mechanical Bowel Preparation

INTERVENTIONS:
Drug: No Mechanical Bowel Preparation — no enemas or oral laxatives will be given in this group
  Arms: No Mechanical Bowel Preparation
Drug: Mechanical Bowel Preparation — oral laxatives (polyethylenglycol at 100 ml/kg/dose for up to 3 times) and stoma enemas (20mlkgdo of normal saline 3 times a day) will be prescribed
  Other Names: Nulitelly
  Arms: Mechanical Bowel Preparation

SUMMARY:
This study will help determine wether mechanical bowel preparation before a colostomy closure is necessary in pediatric population, in order to avoid surgery related complications (surgical site infection and anastomosis leakage).

Half of the population will go through the mechanical bowel prep before colostomy closure and the other half won´t. Complications rate will be compared among both groups.

DETAILED DESCRIPTION:
Mechanical bowel preparation is based on administering osmotic laxatives and enemas through the stomas, in order to diminish solid stool and bacterial load on the colon prior to a colostomy takedown. This was thought to decrease the surgery related complications.

However mechanical bowel preparation can cause discomfort in patients as well as other complications like hydro electrolyte imbalance.

Studies in adult population have shown that there is not a significant difference in the presence of surgery related complications in patients that received bowel prep and those who did not.

There is not enough evidence in pediatric patients that this affirmation is also true.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who are to be submitted to a colostomy closure

Exclusion Criteria:

* patients with more than 3 abdominal surgeries
* patients with primary or acquired immunodeficiencies (including malnourishment)
* Patients in which the distal intestine is closed in a Hartmann´s pouch

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Surgery Related Complications | up to 30 days
  Presence of surgical site infections according to the Centers for Disease Control classification, Presence of anastomotic leakage

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No